CLINICAL TRIAL: NCT03470285
Title: Diagnostic Value of Multiparametric MR Imaging of Small Solid Renal Tumors (IRMK01)
Brief Title: Multiparametric MRI for Diagnosing Small Renal Tumors
Acronym: IRMK01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2015/40
Record Dates: First submitted 2018-02-26; First posted 2018-03-19 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Renal Cancer
Keywords: Mulitparametric MR Imaging; Small solid renal tumors
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with small solid renal tumor (Other): In addition to the actual workflow for a patient presenting a renal tumor, patients will undergo an additional Multiparametric MR imaging (mpMRI).
  Interventions: Procedure: Multiparametric MR imaging (mpMRI)

INTERVENTIONS:
Procedure: Multiparametric MR imaging (mpMRI) — The main objective of the study is to assess the diagnostic accuracy of mpMRI in small renal tumors. The study characteristics will comply with recommended methods (Quadas, Stard). The population to be included will be representative of patients who would benefit from mpMRI if it is demonstrated to be accurate. In this project, the MR protocol will used the conventional MR sequences either on 1.5 or 3T systems and do not require development. Each center may use their own protocol as long as it includes the mandatory sequences.

SUMMARY:
Renal cell carcinoma represents annually 3-5% of all new cancer diagnoses. To date, the standard of care for small renal masses is partial nephrectomy. However, in the specific setting of small renal masses, 20% of them are benign and surgery results in overtreatment. Non-invasive techniques able to differentiate the inherent characteristics of tumors (nature, aggressiveness) would be useful to offer the most appropriate therapeutic options. Morphological ultrasound or CT imaging appeared limited because of the lack of discriminatory power. Based on the data of retrospective studies, the hypothesis is that multiparametric (mp) MR parameters using chemical shift, diffusion and/or contrast injection techniques may be a reproducible diagnostic test with sufficient diagnostic accuracy to differentiate benign from malignant renal tumors. The originality of this project lies in the opportunity to simultaneously assess the performance of mpMRI in diagnosing renal tumors in a routine clinical practice in 18 centers. In each center, two independent MRI readings performed by two radiologists will be carried out within a short delay and interpreted blind to each other's results or pathological results using a predefined template. A third reading will also be centrally performed by the coordinating center according to similar modality. All clinical, radiological and pathological data will be collected after anonymization in the UroCCR database. These informations are used to adjust the therapeutic decision and selecting patients eligible for nephrectomy, other therapeutic options or monitoring.

DETAILED DESCRIPTION:
Renal cell carcinoma represents annually 3-5% of all new cancer diagnoses. In France, its incidence is about 10,000 cases/year. It has been increasing for the past thirty years, probably related to incidental imaging findings. The average age of diagnosis is 65 years. Although the mortality rate started to decrease, partly due to an earlier diagnosis, the overall survival at 5 years is 63% but significantly higher for localized stages (58% of diagnoses): 90%. To date, the standard of care for small renal masses is partial nephrectomy. However, in the specific setting of small renal masses, 20% of them are benign and surgery results in overtreatment. Moreover, for selected patients with comorbidities and potentially low risk tumors, a surveillance strategy can be offered. No preoperative image based tumor characterization has been validated so far, and the kidney tumor biopsy is currently the only way to rule out patients for overtreatment. However, kidney tumor biopsy is invasive, time-consuming, sometimes inconclusive, especially in case of small size tumors, and its low accuracy in predicting tumor aggressiveness based on the Fuhrman grade was several times reported in the literature. Kidney tumor biopsy results may also be impacted by the intra-tumoral heterogeneity. Thus, non-invasive techniques able to differentiate the inherent characteristics of tumors would be useful to offer the most appropriate therapeutic options. Morphological ultrasound or CT imaging appear limited because of the lack of discriminatory power between the different tumor subtypes. Based on the data of retrospective studies, the hypothesis is that MR parameters using chemical shift, diffusion and/or contrast injection techniques may be a reproducible diagnostic test with sufficient diagnostic accuracy to differentiate benign from malignant tumors and better estimate the tumor aggressiveness. To date, no prospective multi-center study on multiparametric (mp) MR imaging of renal tumors has been reported. Although CT-scan explorations are the standard of care in case of renal tumors, MRI offers several advantages over CT including: improved contrast resolution, functional imaging techniques, and the lack of ionizing radiation, which is of particular significance due to growing concerns over cumulative radiation exposure from multi-phase and repeat CT examinations. In particular, the non-ionizing property of MRI may be critical for patients who undergo repeated screening examinations for renal cell carcinoma including those patients under surveillance. By becoming the reference standard for renal mass imaging in clinical practice, multiparametric MRI may help defining the treatment strategy in a non-invasive fashion, resulting in a better selection of patients eligible for nephrectomy, other therapeutic options or surveillance based on tumor aggressiveness estimate, limiting the costs of care and improving patients' quality of life. The originality of this project lies in the opportunity to simultaneously assess the performances of mpMRI in diagnosing renal tumors in a routine clinical practice. In this context, the research will therefore contribute to the development of practical new technologies, strategies and tools for managing renal tumors. MpMRI will be performed in a time-efficient manner and to provide important information that is not available with standard renal MRI or CT-scan. Critical information provided through mpMRI will be used to adjust the therapeutic decision and more adequately select patients eligible for nephrectomy, other therapeutic options or surveillance. Another innovative aspect of the project is to bring together as teamwork several medical disciplines such as radiology, urology, oncology and pathology. The project has been developed and will be conducted within the framework of the French research network on kidney cancer UroCCR (www.uroccr.fr). INCa has been supporting this multidisciplinary network since 2011 and the web-based shared clinical and biological national database on kidney cancer UroCCR will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18;
* Performance Index ≤ 2 (WHO);
* Non hereditary solid renal tumors;
* Indication of renal surgery or renal biopsy for suspicion of malignancy of the tumor
* Size of renal mass between 1,5 and 4 cm;
* Single Renal mass;
* Discovered incidentally by US and / or CT-scan;
* IRMK01 and UroCCR Informed consents signed.
* Affiliated or beneficiary of French social security
* All women of childbearing potential must have effective contraception from the time of screening until MRI. Acceptable methods of contraception include combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal), progestogen-only hormonal contraception (oral, injectable, implantable) intrauterine device, intrauterine hormonereleasing system, bilateral tubal occlusion, vasectomized partner and sexual abstinence

Exclusion Criteria:

Patent signs of malignancy (metastasis, lymphadenopathy, thrombus ...);

* Cystic lesions according to the Bosniak classification;
* Lesions with macroscopic fat on ultrasound or CT-scan;
* Multiple or bilateral renal tumors;
* Histological evidence available initially;
* History of renal neoplasia whatever the location or family context (Von Hippel Lindau, Bourneville sclerosis);
* Moderate to terminal renal impairment documented (creatinine clearance <30 mL / min according MDRD or CKD-EPI);
* Impossibility to perform MRI :

  * heart pacemakers (especially older types)
  * insulin pumps
  * implanted hearing aidsIRMK01 Version no.3.0 of 28/10/2020 Page 12 of 83
  * neurostimulators
  * intracranial metal clips
  * metallic bodies in the eye
* Contraindication to gadolinium salt.
* Patient's refusal of surgery, biopsy if necessary;
* Minor
* Person deprived of liberty
* Person under trusteeship
* Person under curatorship
* Person under legal guardianship
* Pregnant or nursing women.
* Adults unable to express their consent
* Females of child-bearing potential without a negative pregnancy test prior to MRI exam
* Clinical follow-up not possible for psychological, family, social or geographic reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of multiparametric MR imaging (mpMRI) | For MRI results change from 1 day after urologist consultation up to 75 days, for pathology results change from 75 days after urologist consultation up to 3 months
  Index test will be the result from a dichotomized Likert Scale assessing the level of certainty of the malignant of benign nature as assessed by the radiologist on mpMRI images. The reference standard will be the pathology of the tumor (biopsy or surgery). The main measure of interest is the negative predictive value of a dichotomized Likert scale that is rating the level of certainty of the tumor nature diagnosis, based on mpMRI.

SECONDARY OUTCOMES:
Impact of mpMRI on the clinical management of renal tumors | For MDC 1 up to 45 days after first urologist consultation, for MDC 2 up to 75 days after first urologist consultation
  Comparison between management plan decided during MDC1 before mpMRI and during MDC2 after results from mpMRI.
Inter-observer reproducibility of mpMRI | At inclusion
  Comparison between results on Likert scale obtained from 3 readings. Independent assessments by 2 radiologists from the investigating center blind from each other and 1 central reviewer.
  Likert scale (0, 1, 2, 3 or 4) assessing the level of certainty of the malignant or benign nature of the tumor, as assessed by the radiologist on mpMRI images, after coding each of the detailed MRI parameters.
MR parameters in tumor subgroups based on histological findings | For MRI results between from 1 day after urologist consultation up to 75 days, for pathology results from 75 days after urologist consultation up to 3 months
  MR parameters of each renal tumor subgroups assessed by pathology will be compare.
Conclusion about the aggressiveness of clear cell renal cell carcinoma as assessed either by MR parameters or according to Fuhrman grade | For MRI results between from 1 day after urologist consultation up to 75 days, for pathology results from 75 days after urologist consultation up to 3 months
  Conclusions regarding aggressiveness of clear renal cell carcinoma assessed either by MR parameters or according to Fuhrman grade will be compare.
Occurrence of adverse events up to 6 months after mpMRI, initial surgery, biopsy or ablation | From inclusion up to 6 months
  Occurrence assessment of adverse events following MRI, initial surgery, biopsy or ablation
Ancillary RADIOMICS project will be conducted to validate new applied mathematics tools allowing semi-automatic quantitative evaluation of MR images | For MRI results between from 1 day after urologist consultation up to 75 days. Algorithm results, probably 1 year after the end of the study
  A First step will be to provide a precise definition of the tumor volume and will allow to define a signature of each tumor. A statistical learning algorithm will be run in order to propose for each patient a quantification of the probability of malignancy of the tumor according to demographic data and imaging parameters.

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - APHP - Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - APHP - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHRU Lille, Lille
  - CHU Lyon, Lyon
  - APHM - Hôpital de la Conception, Marseille
  - CHU Nancy, Nancy
  - CHU Nice, Nice
  - APHP - Hôpital Tenon, Paris
  - APHP - Hôpital Necker, Paris
  - APHP - Hôpital Bichat, Paris
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No